CLINICAL TRIAL: NCT07299370
Title: Outcomes of Open vs Closed Reduction in Femoral Neck Fractures Using Dynamic Hip Screw
Brief Title: Open vs Closed Reduction in Femoral Neck Fractures Using Anterolateral vs Direct Lateral Approach
Acronym: FNFs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samer youssef mansour meglaa (Other)
Responsible Party: Sponsor-Investigator, Samer youssef mansour meglaa, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: open vs closed reduction FNFs
Record Dates: First submitted 2025-09-18; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-08

CONDITIONS: Femoral Neck Fractures
Keywords: Watson jones approach
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: Comparison between open and closed reduction of femoral neck fractures
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Open eduction of femoral neck fractures (Experimental): Open reduction Using watson jones approach
  Interventions: Device: Open reduction of femoral neck fractures
- Closed reduction of femoral neck fractures (Experimental): Using direct lateral approach
  Interventions: Procedure: Closed reduction of femoral neck fractures

INTERVENTIONS:
Procedure: Closed reduction of femoral neck fractures — Closed reduction of femoral neck fractures
  Arms: Closed reduction of femoral neck fractures
Device: Open reduction of femoral neck fractures — Open reduction of femoral neck fractuctures
  Arms: Open eduction of femoral neck fractures

SUMMARY:
Outcomes of open vs closed reduction if emoral neck fractures

DETAILED DESCRIPTION:
Outcomes of open vs closed reduction in femoral neck fractures using anterolateral vs direct lateral approach using dynamic hip screws

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* patients of both genders between the ages of 16 to 60 years old and had trauma caused femoral neck fracture.
* patients of both genders with Garden's type three and four femoral neck fractures

Exclusion Criteria:

* patients of both genders below the age of 16 and above 60 years old.
* patients with pathological femoral neck fractures.
* patients with autoimmune diseases like rheumatoid arthritis.
* patients with neglected femoral neck fractures(more than 1 week).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation of reduction quality postoperatively | 6 month
  By measuring :
  * 1- femoral offset
  * 2-Neck-length discrepancy
  * 3 - ante-version angle
  * 4-step-off

SECONDARY OUTCOMES:
Asses patients clinically post operative | 1 year
  Using Harris Hip Score

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghayoumi P, Kandemir U, Morshed S. Evidence based update: open versus closed reduction. Injury. 2015 Mar;46(3):467-73. doi: 10.1016/j.injury.2014.10.011. Epub 2014 Oct 14. PMID 25554424
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30712497/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9709424/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20194320/